CLINICAL TRIAL: NCT03878420
Title: A Double-Masked, Randomized, Sham-Controlled, Parallel Group, Multi-Center Study to Assess the Safety and Efficacy of Photobiomodulation (PBM) in Subjects With Dry Age-Related Macular Degeneration (AMD) (LIGHTSITE II)
Brief Title: Study of Photobiomodulation to Treat Dry Age-Related Macular Degeneration (LIGHTSITE II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiThera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSP003
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: Dry AMD; Photobiomodulation; Visual Acuity; Contrast Sensitivity; Optical Coherence Tomography; Drusen

STUDY DESIGN:
Intervention Model Description: Valeda Light Delivery System
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBM Treatment (Experimental): The Valeda™ Light Delivery System will deliver 590, 660 and 850 nm wavelengths together.
  Interventions: Device: Valeda PBM treatment
- Sham Treatment (Sham Comparator): The Valeda™ Light Delivery System will deliver non-effective treatment of the 590 and 660 nm wavelengths together.
  Interventions: Device: Valeda Sham treatment

INTERVENTIONS:
Device: Valeda PBM treatment — The Valeda Light Delivery System delivers 590, 660 and 850 nm wavelengths of light to the study eye. The Valeda Light Delivery System will treat through the open eyelid with the 590 nm and 850 nm wavelengths together. The 660 nm wavelength will be treated through the closed eyelid.
  Arms: PBM Treatment
Device: Valeda Sham treatment — The sham mode emits an approximate 100x reduction in the highest dose for the 660 nm wavelengths as compared to the treatment mode, producing a slightly duller light. The 850 nm (NIR) wavelength (which is not visible light) is not provided in the sham treatment.
  Arms: Sham Treatment

SUMMARY:
This LIGHTSITE II study is a double-masked, sham-controlled, parallel design, prospective multi-site study for the use of PBM as a treatment for visual impairment in subjects with dry AMD.

DETAILED DESCRIPTION:
This study is a double-masked, sham-controlled, parallel design, prospective multi-site study for the use of PBM as a treatment for visual impairment in subjects with dry AMD. The target enrollment is 96 subjects in up to 10 centers in Europe, randomized at a 1:2 ratio into 2 groups: Sham Treatment (S-1) and PBM Treatment (T-2). Once 96 subjects have been enrolled in the study, if there are less than 144 eyes that qualify for the study, additional subjects will be enrolled until 144 eyes have been included in the study.

S-1 will receive 3 sham treatments per week over 3 to 5 weeks starting at Baseline and starting again at Months 4 and 8. T-2 will receive 3 PBM treatments per week over 3 to 5 weeks starting at Baseline and starting again at Months 4 and 8. Each treatment series will total 9 treatments. Neither the subject nor the study staff will know which treatment the subject has been assigned.

Subjects will receive standard visual outcome measurements including Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA, CSV-1000E contrast sensitivity (CS) and the Radner Reading Test prior to and following each treatment series as well as eye exams, fundus photographs, Heidelberg OCT and FAF imaging and optional Optos Ultra Wide Field (UWF) imaging of the retina at selected time intervals. Subjects will also complete the Visual Function Questionnaire 25 (VFQ-25) at selected time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 50 years of age at Screening visit
* Subjects with ETDRS BCVA letter score of between 50* and 75* (Snellen equivalent of 20/100 to 20/32). *If the subject meets this criterion at the Screening Visit but is outside the letter score by up to two letters at Baseline, the subject may be entered in the study.
* Subjects with a diagnosis of dry AMD as defined by the presence of drusen (regular or reticular pseudodrusen) and/or geographic atrophy (GA) visible on two of the following: color fundus images, OCT and/or Heidelberg FAF
* Able to communicate well with the Investigator and able to understand and comply with the requirements of the study
* Subject is informed of the nature of this study and has provided written informed consent in accordance with institutional, local and national regulatory guidelines

Exclusion Criteria:

* Current or history of neovascular maculopathy that includes any of the following:

  1. Choroidal neovascularization (CNV) defined as pathologic angiogenesis originating from the choroidal vasculature that extends through a defect in Bruch's membrane
  2. Serous and/or hemorrhagic detachment of the neurosensory retina or retinal pigment epithelial (RPE)
  3. Retinal hard exudates (a secondary phenomenon resulting from chronic intravascular leakage)
  4. Subretinal and sub-RPE fibrovascular proliferation
  5. Disciform scar (subretinal fibrosis)
* Presence of center involving GA within the central ETDRS 1 mm diameter at Screening
* Media opacities, including cataracts, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require cataract surgery in the study eye in the next 24 months.
* Posterior capsule opacification, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require surgery in the study eye in the next 24 months
* Invasive eye surgery (e.g. cataract, capsulotomy) on a qualifying eye within three 3 months prior to Screening
* Ocular disorder or disease that partially or completely obstructs the pupil (e.g. posterior synechia in uveitis)
* Visually significant disease in any ocular structure apart from dry AMD (e.g. diabetic macular edema, glaucoma (using >2 eye drop medications, uncontrolled IOP and/or central/paracentral visual field loss), glaucoma surgery, active uveitis, active vitreous disease, intraocular tumor, retinal vascular diseases)
* Has a serious medical illness that will prevent the subject from performing study activities (including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease) or, in the judgement of the Investigator, is likely to require surgical intervention or hospitalization at any point during the study
* Presence of or history of malignancy within the past 5 years other than non-melanoma skin or squamous cell cancer or cervical carcinoma in-situ
* Is non-ambulatory
* Presence or history of known light sensitivity to yellow light, red light, or near infrared radiation (NIR), or if there is a history of light activated CNS disorders (e.g. epilepsy, migraine)
* Use of any photosensitizing agent (e.g. topicals, injectables) within 30 days of treatment without consulting subject's physician
* History of drug, alcohol or substance abuse within 3 months prior to Screening
* Has received an investigational drug or treatment with an investigational device within 3 months prior to Screening
* If on any anti-oxidant or vitamin Age-Related Eye Disease Study (AREDS) supplement for dry AMD, has not been stabilized for a minimum of 1 month prior to Screening. Subjects are considered to be stable if they are taking the AREDS supplements consistently as prescribed by their treating doctor.
* Has received Low Vision Rehab/Therapy within 30 days prior to Screening or intends to receive during the study
* In the opinion of the Investigator, is unlikely to comply with the study protocol

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | Month 9
  The primary efficacy endpoint will be the change in BCVA from Baseline to Month 9 as assessed using the ETDRS BCVA chart.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | Month 9
  The first of the secondary analyses will test the difference between the sham-treated and PBM-treated subjects in mean change from baseline (pre-treatment) to Month 9 in BCVA.
Contrast Sensitivity | Month 9
  The second of the secondary analyses will test the difference between the sham-treated and PBM-treated subjects in mean change from baseline (pre-treatment) to Month 9 in contrast sensitivity at 18 cycles/degree (CPD).
Impact on Central Drusen Volume by OCT | Month 10
  The analyses will first examine change from the screening visit in central Drusen volume
Impact on Central Drusen Thickness by OCT | Month 10
  The analyses will then examine change from the screening visit in central Drusen Thickness

CONTACTS AND LOCATIONS:
Locations (8):
- Institut ophtalmologique de l'Ouest- Clinique jules VERNE, Nantes, France
- Germany (3):
  - Universitätsklinikum Freiburg- Klinik für Augenheilkunde, Freiburg im Breisgau
  - Klinik fur Ophthalmologie, Universitatsklinikum Schleswig-Holstein, Kiel
  - Universitaetsmedizin Mainz- Augenklinik, Mainz
- Osprdalr San Raffaele, Milan, Italy
- Institut Català de Retina, Barcelona, Spain
- United Kingdom (2):
  - James Paget University, Great Yarmouth
  - Peterborough City Hospital, Peterborough

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Burton B, Parodi MB, Jurgens I, Zanlonghi X, Hornan D, Roider J, Lorenz K, Munk MR, Croissant CL, Tedford SE, Walker M, Ruckert R, Tedford CE. LIGHTSITE II Randomized Multicenter Trial: Evaluation of Multiwavelength Photobiomodulation in Non-exudative Age-Related Macular Degeneration. Ophthalmol Ther. 2023 Apr;12(2):953-968. doi: 10.1007/s40123-022-00640-6. Epub 2023 Jan 2. PMID 36588113